CLINICAL TRIAL: NCT03771976
Title: Risk of Cesarean Section and Perinatal Complications in Primiparous Women Over 35 Years of Age. A Retrospective Cohort Study.
Brief Title: Risk of Cesarean Section in Primiparous Women Over 35 Years of Age.
Status: Completed | Type: Observational
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Chairman of Research - Saint Thomas Maternity Hospital, Saint Thomas Hospital, Panama
Other Study IDs: MHST-2014-05
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Pregnancy Complications
Keywords: Older women (>35 years of age); Primipara; Cesarean section
MeSH Terms: conditions — Pregnancy Complications | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Over 35 years of age: Primiparous women over 35 years of age.
  Interventions: Procedure: Cesarean section; Procedure: No cesarean section
- Between 20-34 years of age: Primiparous women between 20 and 34 years of age.
  Interventions: Procedure: Cesarean section; Procedure: No cesarean section

INTERVENTIONS:
Procedure: Cesarean section — Risk of cesarean section between the cohorts
Procedure: No cesarean section — Vaginal birth rate between the cohorts

SUMMARY:
The investigators reviewed Saint Thomas Maternity Hospital's database during a 5 year period and compared two cohorts of patients (primiparous women over 35 years of age and primiparous woman between 20 and 34 years of age). The objective was to determine the risk of cesarean section and other perinatal complications between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Primiparous women.
* Birth after 22 weeks and neonatal weight > 501g.

Exclusion Criteria:

* Multiparity.
* Birth before 22 weeks or neonatal weight < 500g.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primiparous women, between 22 and 42 weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Risk of cesarean section | 5 years
  Rate of cesarean sections (birth by cesarean section), independent of the reason.

SECONDARY OUTCOMES:
Perinatal complications | 5 years
  Any combination of perinatal complications (Stillbirth, low apgar score) between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas H, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data. Just the final results.